CLINICAL TRIAL: NCT04155489
Title: The Impact of Perioperative Restrictive Transfusion on Postoperative Cognitive Dysfunction in Elderly Patients Undergoing Spine Surgery
Brief Title: The Impact of Perioperative Transfusion on Postoperative Cognitive Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Yon Hee Shim, Professor,Department of Anesthesiology and Pain Medicine, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3-2019-0271
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: POCD; Anemia; Transfusion
MeSH Terms: conditions — Anemia | interventions — Blood Transfusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- restrictive (Active Comparator): In the restrictive blood transfusion group, if the hemoglobin value is less than 8 g /dL or if there are suspected symptoms of anemia such as dizziness or chest pain, headache, low on energy, blood transfusion is started.
  Interventions: Procedure: blood transfusion
- Liberal (Experimental): In the liberal transfusion group, If the hemoglobin value is less than 10 g /dL, blood transfusions begin.
  Interventions: Procedure: blood transfusion

INTERVENTIONS:
Procedure: blood transfusion — In the restrictive blood transfusion group, if the hemoglobin value is less than 8 g /dL or if there are suspected symptoms of anemia such as dizziness or chest pain, headache, low on energy, blood transfusion is started. in the liberal transfusion group, If the hemoglobin value is less than 10 g /dL, blood transfusions begin.

SUMMARY:
Although blood transfusion is a representative treatment for acute anemia due to blood loss during surgery, it is also a powerful risk factor for postoperative cognitive dysfunction.

'Restrictive transfusion', which transfusions minimal red blood cells, is not only useful for conserving limited blood resources, but also does not worsen prognosis or mortality after surgery. Research has also been reported that severe restrictive transfusion has improved prognosis and mortality.

However, anemia is also one of the risk factors for postoperative complications, including neurocognitive impairment, it is still controversial how much anemia should be allowed in elderly people who are sensitive to ischemia or heart disease.

The purpose of this study is to determine whether the restrictive transfusion policy reduces the frequency of postoperative cognitive dysfunction than the liberal transfusion policy in patients aged 65 years or older who undergo lumbar interbody fusion.

Restrictive transfusion strategy (which initiates transfusion when hemoglobin level is less than 8 g / dL during perioperative period) // liberal transfusion strategy (which initiates transfusion when hemoglobin level is less than 10 g / dL during perioperative period)

DETAILED DESCRIPTION:
The Aim of this study was to compare the frequency of postoperative cognitive dysfunction diagnosed 7 days after surgery between two groups.

K-MOCA (Korean-Montreal Cognitive Assessment) is used to evaluate cognitive dysfunction. In addition, plasma inflammatory markers (CRP, IL-6) and GFAP reflecting brain damage were measured before and after surgery to determine whether brain injury caused by systemic inflammatory response is associated with cognitive dysfunction

ELIGIBILITY:
Inclusion Criteria:

* Patients 65 years of age or older who receive more than two levels of lumbar interbody fusion

Exclusion Criteria:

* If patients have anemia (Hb is less than 13 g / dL for men and less than 12 g / dL for women)
* Those who cannot read the agreement (illiteracy, foreigner, etc.)
* Have a history of taking medication for mental illness
* Communication disorders due to neurological diseases (dementia, stroke, seizures, etc.)
* Less than 23 points on K-MoCA test
* When fluid loading and volulyte are difficult due to kidney disease
* Limited blood transfusion due to heart disease
* Refusal of blood transfusions (religious reasons, etc.)
* patients who have received a blood transfusion within 6 weeks prior to surgery
* If continuous observation is impossible after surgery
* Emergency surgery

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2020-01-08 (Actual); Primary Completion 2024-10-14 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Comparing the frequency of post-operative cognitive dysfunction diagnosed on the 7th day after surgery | 7th day after surgery (POD 7)
  On the day before the surgery and the seventh day after the surgery, the patient scan K-MOCA (Korean-Montreal Cognitive Assessment). If the difference between the preoperative test results and the post-operative test results is RCI (Reliable Change Index) <-1.96, it is determined that cognitive dysfunction occurred.

CONTACTS AND LOCATIONS:
Overall Officials: Yonhee Shim, Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

REFERENCES:
- [Background] Behrends M, DePalma G, Sands L, Leung J. Association between intraoperative blood transfusions and early postoperative delirium in older adults. J Am Geriatr Soc. 2013 Mar;61(3):365-70. doi: 10.1111/jgs.12143. PMID 23496244
- [Background] Chen QH, Wang HL, Liu L, Shao J, Yu J, Zheng RQ. Effects of restrictive red blood cell transfusion on the prognoses of adult patients undergoing cardiac surgery: a meta-analysis of randomized controlled trials. Crit Care. 2018 May 31;22(1):142. doi: 10.1186/s13054-018-2062-5. PMID 29848364
- [Background] Deiner S, Silverstein JH. Postoperative delirium and cognitive dysfunction. Br J Anaesth. 2009 Dec;103 Suppl 1(Suppl 1):i41-46. doi: 10.1093/bja/aep291. PMID 20007989
- [Background] Fan YX, Liu FF, Jia M, Yang JJ, Shen JC, Zhu GM, Zhu SH, Li WY, Yang JJ, Ji MH. Comparison of restrictive and liberal transfusion strategy on postoperative delirium in aged patients following total hip replacement: a preliminary study. Arch Gerontol Geriatr. 2014 Jul-Aug;59(1):181-5. doi: 10.1016/j.archger.2014.03.009. Epub 2014 Mar 29. PMID 24745810
- [Background] Fusaro MV, Nielsen ND, Nielsen A, Fontaine MJ, Hess JR, Reed RM, DeLisle S, Netzer G. Restrictive versus liberal red blood cell transfusion strategy after hip surgery: a decision model analysis of healthcare costs. Transfusion. 2017 Feb;57(2):357-366. doi: 10.1111/trf.13936. Epub 2016 Dec 26. PMID 28019009
- [Background] Hudetz JA, Gandhi SD, Iqbal Z, Patterson KM, Pagel PS. Elevated postoperative inflammatory biomarkers are associated with short- and medium-term cognitive dysfunction after coronary artery surgery. J Anesth. 2011 Feb;25(1):1-9. doi: 10.1007/s00540-010-1042-y. PMID 21061037